CLINICAL TRIAL: NCT04192370
Title: A Single-arm, Open-label Feasibility Pilot of Cannabidiol as an Adjunct to Sublingual Buprenorphine on Cue-induced Cravings Among Individuals With Opioid Use Disorder
Brief Title: Cannabidiol Use to Reduce Cravings in Individuals With Opioid Use Disorder on Buprenorphine
Acronym: CURB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P003384
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cannabidiol (Experimental): As this is a single-arm, open-label study, all subjects will receive the interventional arm, specifically 600mg of oral cannabidiol once daily for 3 consecutive days.
  Interventions: Drug: Cannabidiol 600mg

INTERVENTIONS:
Drug: Cannabidiol 600mg — All subjects will receive 600mg of oral cannabidiol for 3 days in an open-label fashion. Cannabidiol will be provided using Epidiolex™ oral solution 100mg/mL, and the drug will be procured by the Brigham and Women's Hospital (BWH) Investigational Drug Services (IDS) pharmacy. The first dose will be administered at the BWH Center for Clinical Investigation, while doses 2 and 3 will be self-administrated at home. The CBD will be repacked in pre-drawn syringes for the subjects to self-administer at home.
  Other Names: CBD; Epidiolex

SUMMARY:
The purpose of this week-long study is to determine the impact of cannabidiol on cue-induced cravings among individuals with opioid use disorder who are stable on sublingual buprenorphine treatment.

DETAILED DESCRIPTION:
Studies have indicated that medication treatment for opioid use disorder (OUD) with buprenorphine, methadone, or extended-release naltrexone reduces the risk for overdose by 70%. However, treatment dropout rates remain unacceptably high, with approximately 50% of patients discontinuing treatment 6 months after initiation. There is a substantial body of research indicating that high rates of treatment discontinuation are due to the emergence of intense cravings to use illicit opioids in response to cues - which are reminders of the drug such as drug paraphernalia. Much of the research so far in improving treatment retention on medications for OUD have focused on helping patients learn how to avoid triggers and to manage their cravings if they do emerge, and psychosocial treatments as adjuncts to medications has similarly not been as helpful as hoped. As such, there is a critical need to identify novel strategies that will improve retention in medical treatment for OUD, and cannabidiol (CBD) has emerged as a possible adjunct to OUD treatment, as it appears to target brain regions that mediate cue-induced cravings. Two studies so far have shown that CBD reduces cue-induced cravings for abstinent individuals with OUD not taking any medications, but the impact of CBD on cue-induced cravings among individuals stabilized on buprenorphine is not known.

Given that long-term medication treatment remains the gold-standard approach, a critical question that remains unanswered is whether CBD can be used as an adjunct to buprenorphine treatment to reduce cue-induced cravings. As such, the purpose of this week-long open-label feasibility pilot is to determine the impact of cannabidiol on cue-induced cravings among individuals with opioid use disorder who are stable on sublingual buprenorphine treatment. Patients with OUD currently receiving treatment with sublingual buprenorphine will be eligible to enroll. The cue-induced cravings assessment will be conducted before and after the CBD administration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) opioid use disorder, severe
* Currently in treatment with methadone or buprenorphine

Exclusion Criteria:

* Requiring level of care higher than outpatient treatment for alcohol, sedative/hypnotics, or stimulants
* Any current mood episode requiring level of care higher than outpatient treatment
* History of psychotic disorder or bipolar disorder
* Currently pregnant
* Hepatic liver enzymes greater than 3x upper normal limit
* Hypersensitivity to cannabinoids or sesame oil (cannabidiol solution comes in sesame oil emulsion)
* Currently taking any medications with known significant pharmacokinetic interactions with CBD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki J, Martin B, Prostko S, Chai PR, Weiss RD. Cannabidiol Effect on Cue-Induced Craving for Individuals with Opioid Use Disorder Treated with Buprenorphine: A Small Proof-of-Concept Open-Label Study. Integr Med Rep. 2022 Aug 1;1(1):157-163. doi: 10.1089/imr.2022.0070. Epub 2022 Aug 26. PMID 36105269

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol
Started | 8
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: The number of participants at baseline is 7 instead of 8 because one patient who was consented and enrolled according to the protocol left the study site before any baseline measures were able to be collected and decided to withdraw from the study.
Arm/Group | Cannabidiol
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.86 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Cue-induced Cravings and Anxiety After 3 Days of Cannabidiol Administration
Description: Change in cue-induced cravings and anxiety measured before and after 3 days of cannabidiol administration. Subjects will use the Cue-Induced Opioid Craving and Anxiety Scales to note their responses using a visual analog scale of 0 to 10, 0 being "not at all" and 10 being "extremely." Higher scores thus mean a "worse" outcome (i.e. more intense cravings/anxiety).
Time Frame: pre-exposure (Visit 2, which is day 2 of the 5-day study) and post-exposure (Visit 3, which is day 5 of the 5-day study)
Population: Individuals with opioid use disorder who are currently receiving buprenorphine for treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol
Number analyzed (Participants) | 5
score on a scale
  Cannabidiol | 3.2 (.8)
  Pre-CBD | 0.4 (0.5)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse Events were monitored/assessed, but none observed.
Arm/Group | Cannabidiol
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04192370/Prot_SAP_000.pdf